CLINICAL TRIAL: NCT05715359
Title: Standardized Osteotomy Guides for Free Flap Reconstruction of Continuous Defects of the Jaws - a Simplified Method
Status: Enrolling by invitation | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Martin Bengtsson, DDS, PhD, Consultant Oral and Maxillofacial Surgeon, Lund University Hospital
Other Study IDs: Standardized osteotomy guide
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Oral Surgical Procedures; Surgery, Oral; Mandibular Reconstruction
Keywords: Maxillofacial; Reconstruction; Osteotomy; Maxilla; Mandible
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reconstruction of jaws.: Patients treated with free tissue transfer reconstruction of the jaws.
  Interventions: Procedure: Reconstruction

INTERVENTIONS:
Procedure: Reconstruction — Standardized template for reconstruction of continious defects of the jaws.

SUMMARY:
The aim of the present project is to evaluate the outcome from reconstruction of the jaws, with a standardized simplified technique, after a continuous defect.

The primary objective is to measure recurrence of the tumour is present as a marking for insufficient resection margins. Secondary objectives are measures of survival of transplanted tissues, registered complications at follow-up and measures of healing between segments of transplanted bone (bone bridging).

DETAILED DESCRIPTION:
Subjects The participants in this retrospective survey were consecutive head- and neck malignancy patients referred 2002-2021 to Skåne University Hospital, Lund, Sweden with an osseous proximity or malignancy. The treatment consisted of combined surgical resection and radiotherapy. Patients will be identified through the use of ICD-coding. All patients included underwent a primary functional and aesthetical reconstruction of continuous defects of the jaws with free vascularized tissue transfer adopted to the area of resection with the aid of a standardized osteotomy guide. The subjects eligible for inclusion in this project should present at least 1-year postoperative follow-up.

Patients eligible for inclusion will be notified in newspaper announcement. One announcement in a national newspaper and one announcement in the member newspaper of the Association for oral and neck cancer patients. Patients that are not agreeing to take part in this project are expected to declare this to the primary investigator. A drop-out analysis will be performed on 30 of the not included subjects according to age and gender.

Surgical Method Reconstruction of resected osseous anatomy was performed on the same occasion as tumour resection. Increased resection margins were decided after marginal intraoperative frozen autopsies. The reconstruction was performed aiming for maximal function with the best possible aesthetic outcome. All patients were initially planned to finalize the reconstructive phase with a dental rehabilitation of dentition lost during the oncological treatment. When applicable, a full dental rehabilitation was performed at least 12 months after resection.

Surgically, a non-customized template with dimensions taken from The Brånemark Novum® concept was used. Hence, the in-house template and cutting guide design was based upon a mean dimension of the size and form in a fully-grown individual. A sectioning of the transplant into three pieces, one frontal and two lateral, for reconstruction of the mandibular body was used as the base for the design. The angle between the segments was designed into aslant of thirty degrees.

The template and cutting guide were initially designed for mandibular reconstruction with an osseo-musculo-cuttaneous vascularized fibula graft. With time, the design was also suitable and used for reconstruction of maxillary and midface reconstruction and in cases with other flaps, like the tip and lateral rim of scapula.

Gradually, the cutting guide for the mandibular body angle was also usable when reconstructing the angle between the body and ramus of the mandible. Further, the angle of the guide was also found to be usable for a reconstruction of the maxillary base at the level suitable to a prosthetic reconstruction of the alveolar process and maxillary dentition to fit a mandibular dentition.

From a biomechanical aspect, the transplant was fixated to the anatomical region with a load sharing principle, meaning osteosynthesis not overbridging the segments but only connecting them. Thus, the transplanted bone was partly loaded to catalyse the osteogenesis. For the same reason, the remaining osseous tissues were, in accordance to a previous study, handled predominately without stripping of the periosteum.

All subjects were treated with postoperative RT, having implant supported dental rehabilitation to be performed in radiated tissues. When applicable, dental rehabilitation begun no earlier than 1 year after tumour resection and after radiographic verification of bone bridging between transplanted bone segments. To improve the healing capacity, hyperbaric oxygene therapy (HBO) was performed at a daily basis four weeks before and two weeks after implant insertion. Ten days per oral antibiotic was given with start two days prior to implant insertion. Implants were loaded six months after insertion.

Variables and data collection methods Registrations from patient journals and radiographs will include the following variables

1. Survival (patient).
2. Recurrent tumour.
3. Complications (including tissue survival).
4. Function.
5. Healing of bone segment (bone bridging).
6. Age.
7. Gender.
8. Time since tumour resection.
9. Level of rehabilitation (e.g. dental).
10. Jaw movements (range).
11. Pain.
12. Any problems with per oral nutrition.

The recordings will be collected in an Excel document and the patients will be coded. Identification possibility is limited to the identification of eligible subjects. After that the subjects will be coded and not possible to identify except with the coding list. The coding list will be kept by the primary investigator in a secure, IT-protected server within the Region Skåne. Data analysis and handling will be performed by the investigators on a material not possible to identify individuals in. The results will be presented in a group level without possibility to identify individuals.

Statistical analysis The sample constitutes of a total inclusion from a cohort limited in time, department and treatment method. The project is designed as an observational trial without a group for comparison. Thus, a power-analysis has not been possible to perform, neither is it valued necessary for this project.

Simple statistical analysis including mean, standard deviation and range will be used.

The limit for statistical significance will be set to p<0.05. A two-sided p-value will be used.

ELIGIBILITY:
Inclusion Criteria:

Treated at Skåne University Hospital, Lund, Sweden between 2002-2021 with reconstruction of the jaws using a standardized osteotomy guide.

Exclusion Criteria:

Less than one year follow-up.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated at Skåne University Hospital, Lund, Sweden between 2002-2021 with reconstruction of the jaws using a standardized osteotomy guide.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Reccurence of tumour. | At least one year follow-up after resection.
  Reccurent tumour meaning not radical resection margins

SECONDARY OUTCOMES:
Tissue transfer survival | At least one year follow-up after resection.
  Survival of tissue transfer meaning vital structures remaining in reconstructed region.
Oral function | At least one year follow-up after resection.
  Oral function meaning ability to breathe, chew, swallow and speek.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bengtsson, DDS, PhD, Principal Investigator — Lund University Hospital
Locations (1):
- Dept Oral and Maxillofacial Surgery, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No